CLINICAL TRIAL: NCT01706510
Title: A Single Center, Randomized, Open Label, Multiple Dose, Crossover Study of the Antiplatelet Effects of Ticagrelor Versus Clopidogrel in American Indian Patients With Stable Coronary Artery Disease
Brief Title: Antiplatelet Effects of Ticagrelor Versus Clopidogrel in American Indian Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rapid City Regional Hospital, Inc (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0076
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease
Keywords: Clopidogrel; Ticagrelor; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Platelet Aggregation Inhibitors; Hematologic Agents; Therapeutic Uses; Pharmacologic Actions; Purinergic P2Y Receptor Antagonists; Purinergic P2 Receptor Antagonists; Purinergic Antagonists; Purinergic Agents; Physiological Effects of Drugs
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 180 mg loading dose followed by 90 mg bid for 7 days ± 2 days
  Interventions: Drug: Ticagrelor; Drug: Clopidogrel
- Clopidogrel (Active Comparator): Clopidogrel 600 mg Loading Dose followed by 75 mg Daily for 7 days ± 2 days
  Interventions: Drug: Ticagrelor; Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 180 mg loading dose followed by 90 mg bid for 7 days ± 2 days
  Other Names: Brand Name: Brilinta
Drug: Clopidogrel — Clopidogrel 600 mg loading dose followed by 75 mg Daily for 7 days ± 2 days
  Other Names: Brand Name: Plavix

SUMMARY:
Assess the pharmacodynamic effect of ticagrelor vs. Clopidogrel in American Indian patients with stable coronary artery disease.

DETAILED DESCRIPTION:
A Single Center, Randomized, Open Label, Multiple Dose, Crossover Study of the Antiplatelet Effects of Ticagrelor Versus Clopidogrel in American Indian Patients With Stable Coronary Artery Disease

ELIGIBILITY:
Inclusion Criteria:

* Documented stable CAD fulfilling any of the following, and taking 81mg ASA daily treatment:
* Females must be post menopausal for at least one year or surgically sterile for at least 6 months and negative urine pregnancy test
* Self-identified as American Indian
* Genetic Inclusion Criteria: must sign the informed consent for genetic and biological sample banking.

Exclusion Criteria:

* Any indication for oral anticoagulant or dual antiplatelet treatment
* Concomitant therapy with strong CYP3A inhibitors, CYP3A substrates with narrow therapeutic index, or strong CYP3A inducers within 14 days and during study treatment and during:
* Increased bleeding risk including:
* Diabetic patients with HbAlC > 10% at screening
* Contraindication to clopidogrel, ASA, or ticagrelor - A history of alcohol and/or substance abuse that could interfere with conduct of the trial
* Patients requiring dialysis
* Patients scheduled for revascularization (e.g., PCI, CABG) during the study period
* Any acute or chronic unstable condition in the past 30 days
* Known active or recurrent hepatic disorder
* Patients who had ACS or stent placed within 12 months of screening
* History of Uric Acid nephropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Compare ticagrelor's versus clopidogrel's inhibition of the P2Y12 receptor as measured by the decrease in P2Y12 Reaction Units (PRU) using VerifyNow TM. | At 2 hour time point after loading dose

SECONDARY OUTCOMES:
Compare the decrease of P2Y12 Reaction Units (PRU) by VerifyNow TM from ticagrelor and clopidogrel. | 0.5 and 8 hour time points after loading dose
Compare the decrease in P2Y l2 Reaction Units (PRU) by VerifyNow™ from ticagrelor's and clopidogrel's morning dose on Day 7 | At the 2, 8, and 24 hours after the last dose
To evaluate and compare the pharmacodynamic effects, measured by the vasodilator-stimulated phosphoprotein (VASP) assay (platelet reactivity index [PRI]), in all subjects | Day1: pre-dose, 0.5, 2, and 8 hours post loading dose Day 7: pre-dose, 2 and 8 hours post dose Day 8: 24 hours post final dose
Assess and to compare the percentage of subjects with High on-treatment Platelet Reactivity (HPR) at all time points after randomized study treatment. | Day 1: Pre-dose, 0.5, 2 and 8 hours post loading dose Day 7: pre-dose, 2 and 8 hours post dose Day 8: 24 hours after final dose
  The High on-treatment Platelet Reactivity will be defined in accordance with the following platelet inhibition level cut-off.
  * > 208 PRU by the VerifyNow P2Y12 assay
  * > 230 PRU by the VerifyNow P2Y12 assay
  * > 50% PRI by the VASP assay

OTHER OUTCOMES:
CYP2C19 genotyping to identifying the wild-type CYP2C19 allele (*1), and characterize common alleles known to effect the metabolism of clopidogrel (*2, *3, *4,*5,*6,*7,*8 responsible for poor metabolism and *17 allele responsible for rapid metabolism). | One time-point

CONTACTS AND LOCATIONS:
Overall Officials: James S Walder, MD, Principal Investigator — Rapid City Regional Hospital
Locations (1):
- Regional Heart Doctors/Black Hills Cardiovascular Research, Rapid City, South Dakota, United States